CLINICAL TRIAL: NCT04013334
Title: A Phase 2, Open-Label, Single-Center Study of MTG201 in Combination With Nivolumab in Patients With Relapsed Malignant Pleural Mesothelioma
Brief Title: MTG201 Plus Nivolumab in Patients With Relapsed Pleural Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Momotaro-Gene Inc. (Industry)
Collaborators: Baylor College of Medicine (Other); Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTG201-MPM-001
Record Dates: First submitted 2019-05-24; First posted 2019-07-09 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Single arm, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MTG201 plus Nivolumab (Experimental): Single arm, open-label, patients receive both MTG201 and nivolumab
  Interventions: Drug: MTG201; Drug: Nivolumab Injection [Opdivo]

INTERVENTIONS:
Drug: MTG201 — MTG201, 3 x 10E12 vp delivered by intratumoral injection on days 1, 8, 22 and 50
  Other Names: Ad-SGE-REIC/Dkk-3
Drug: Nivolumab Injection [Opdivo] — Nivolumab 480 mg by IV infusion every 4 weeks
  Other Names: Opdivo

SUMMARY:
Twelve patients with relapsed malignant pleural mesothelioma will be treated with intratumoral injections of MTG201, a replication incompetent adenovirus, modified by the insertion of the reduced expression in immortalized cells (REIC)/Dikkopf (Dkk)-3 gene, on Days 1, 8, 22, and 50. Patients will also receive every 4 weekly intravenous infusions of nivolumab, 480 mg, starting on Day 2. Safety and anti-tumor activity will be monitored at regular intervals throughout the study.

DETAILED DESCRIPTION:
This is a study of the efficacy and safety of MTG201 given by intratumoral injection to patients with malignant pleural mesothelioma who have failed front line chemotherapy. Patients will also receive IV infusions of nivolumab every 4 weeks. MTG201 is a replication incompetent adenovirus into which the gene for REIC/Dkk-3 has been inserted. The insertion of this gene has been shown to endow the adenovirus with anti-tumor activity and to result in enhanced anti-tumor immunity.

MTG201, 3 x 10E12 vp, will be given by intratumoral injection on days 1, 8, 22 and 50. Nivolumab, 480 mg, will be given by IV infusion every 4 weeks until progression. Efficacy will be assessed by CT scans at 4 and 12 weeks, then every 3 months. Safety will be assessed by reported adverse events, periodic laboratory assessments, physical exams, vital signs. The pharmacokinetics and pharmacodynamics of MTG201 will be assessed periodically. Tumor biopsy will be obtained on Days 1, 8 and 50 prior to MTG201 administration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic pleural mesothelioma
* Failed one prior treatment regimen including cisplatin-based chemotherapy
* Eastern cooperative oncology group (ECOG) performance status; 0,1
* Adequate organ function
* Measurable disease per RECIST

Exclusion Criteria:

* Candidate for surgical resection
* has active autoimmune disease, primary or acquired immunodeficiency
* significant cardiovascular disease
* has active interstitial lung disease
* has active infection or HIV, hepatitis B or C
* previous anti-PD-1, PD-L1 or CTLA-4 inhibitor immunotherapy
* other clinical significant disorder that could affect conduct of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 months-2 years
  Percentage of subjects with complete or partial response

SECONDARY OUTCOMES:
duration of response (DUR) | up to 2 years
  measured from first observation of response to disease progression
progression free survival (PFS) | up to 2 years
  measured from start of study to date of progression or death

OTHER OUTCOMES:
Incidence of adverse events | up to 2 years
  description of adverse events by frequency, severity and causality
change from baseline in liver transaminases | up to 2 years
  changes in liver transaminases from prior to first study drug treatment to various timepoints throughout the treatment and follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Burt, MD, Principal Investigator — Baylor College of Medicine Thoracic Surgery
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No